CLINICAL TRIAL: NCT02316106
Title: A Randomized Phase 2 Trial to Evaluate Three Daratumumab Dose Schedules in Smoldering Multiple Myeloma
Brief Title: A Study to Evaluate 3 Dose Schedules of Daratumumab in Participants With Smoldering Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR106449; 54767414SMM2001 (Other: Janssen Research & Development, LLC); 2014-005139-14 (EudraCT Number)
Record Dates: First submitted 2014-12-10; First posted 2014-12-12 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
Keywords: Smoldering multiple myeloma (SMM); Daratumumab
MeSH Terms: conditions — Multiple Myeloma; Smoldering Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Long Intense) (Experimental)
  Interventions: Drug: daratumumab
- Arm B (Intermediate) (Experimental)
  Interventions: Drug: daratumumab
- Arm C (Short Intense) (Experimental)
  Interventions: Drug: daratumumab

INTERVENTIONS:
Drug: daratumumab — 16 mg/kg administered by intravenous (IV) infusion once every week in Cycle 1, every other week in Cycle 2 and Cycle 3, every 4 weeks in Cycle 4 to Cycle 7, and from Cycle 8 to Cycle 20 on Day 1 of each cycle. If, as per investigator discretion, there is a positive benefit/risk ratio, absence of Grade greater than or equal to (>=) 3 treatment related toxicity, and at least stable disease has been achieved, treatment can be extended and given every 8 weeks after Cycle 20. For participants participating in treatment extension, the duration of infusion may be shortened to a 90-minute infusion or can switch to daratumumab 1800mg subcutaneous (Q8w).
  Arms: Arm A (Long Intense)
Drug: daratumumab — 16 mg/kg administered by IV infusion once every week in Cycle 1, and then on Day 1 of each cycle from Cycle 2 to Cycle 20, and every 8 weeks after Cycle 20. If, as per investigator discretion, there is a positive benefit/risk ratio, absence of Grade greater than or equal to (>=) 3 treatment related toxicity, and at least stable disease has been achieved, treatment can be extended and given every 8 weeks after Cycle 20. For participants participating in treatment extension, the duration of infusion may be shortened to a 90-minute infusion or can switch to daratumumab 1800mg subcutaneous (Q8w).
  Arms: Arm B (Intermediate)
Drug: daratumumab — 16 mg/kg administered by IV infusion once every week in Cycle 1 only. Treatment cycles are 8 weeks in length.
  Arms: Arm C (Short Intense)

SUMMARY:
The purpose of this study is to evaluate three daratumumab dose schedules in participants with Smoldering Multiple Myeloma.

DETAILED DESCRIPTION:
This is a randomized, open-label (identity of assigned treatment will be known to participants and study staff), 3-arm (3 treatment groups), multicenter study of daratumumab in participants diagnosed with intermediate or high-risk Smoldering Multiple Myeloma (SMM [ie, early disease without any symptoms]). Participants will be randomized (assigned by chance) to one of 3 treatment groups (arm A [long intense], arm B [intermediate] and arm C [short intense]) to receive daratumumab. Each treatment group will investigate 1 of 3 dosing schedules of daratumumab. The study will include a 28-Day Screening Phase, a Treatment Phase of 1 to 20 treatment cycles (each cycle is 8 weeks in duration for total period of 8 to 160 weeks), and a Follow up Phase of 4-weeks from the last dose of study drug. For participants in Arm A (long intense) and Arm B (intermediate), there is a possibility to extend treatment with IV daratumumab (Q8W) after the end of Cycle 20 if, as per investigator discretion, there is a positive benefit/risk ratio, absence of Grade >=3 treatment related toxicity, and at least stable disease has been achieved. For participants participating in treatment extension, the duration of infusion may be shortened to a 90-minute infusion or can switch to daratumumab 1800mg subcutaneous (Q8w). The Follow-up Phase will continue until death, lost to follow up, consent withdrawal, or study end, whichever occurs first. The end of the study will occur approximately 7 years after the last participant enrolled receives a first dose of study drug. 'Disease assessment will be performed locally per Standard of Care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of smoldering multiple myeloma (SMM) for less than 5 years
* Have a confirmed diagnosis of intermediate or high-risk SMM, and an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.

Exclusion Criteria:

* Active multiple myeloma,requiring treatment as defined by the study protocol
* Primary systemic AL (immunoglobulin light chain) amyloidosis
* Prior or concurrent exposure to any of the following: approved or investigational treatments for SMM or/and multiple myeloma, daratumumab or other anti CD-38 therapies, treatment with corticosteroids with a dose greater than (>) 10 milligram (mg) prednisone per day or equivalent and bone-protecting agents (eg, bisphosphonates, denosumab) or are only allowed if given in a stable dose and for a nonmalignant condition, or received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 4 weeks before Cycle 1, Day 1
* History of malignancy (other than SMM) within 3 years before the date of randomization, except for the following if treated and not active: basal cell or nonmetastatic squamous cell carcinoma of the skin, cervical carcinoma in situ, ductal carcinoma in situ of breast, or International Federation of Gynecology and Obstetrics (FIGO) Stage 1 carcinoma of the cervix
* Known chronic obstructive pulmonary disease (COPD) OR moderate or severe persistent asthma within the past 2 years
* Any concurrent medical or psychiatric condition or disease (eg, autoimmune disease, active systemic disease, myelodysplasia) that is likely to interfere with the study procedures or results, or that in the opinion of the investigator, would constitute a hazard for participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
The percentage of participants who achieve a complete response (CR) | Up to 7 years
  CR, defined having negative immunofixation on the serum and urine, and <5% plasma cells (PCs) in bone marrow.
The percentage of participants that have an event (disease progression or death) per patient-year | Up to 7 years

SECONDARY OUTCOMES:
The percentage of participants who are minimal residual disease (MRD) negative | Up to 7 years
Time to next treatment (TNT) | Up to 7 years
  TNT, defined as the time from the date of randomization to the date of the first subsequent multiple myeloma treatment.
The percentage of participants who achieve a Complete Response (CR) or a Partial Response (PR) | Up to 7 years
  See definition of CR above. PR, defined as >=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to <200 mg/24 hours.
The median time of progression free survival (PFS) | Up to 7 years
  PFS is defined as time from date of randomization to date of initial documented disease progression (PD) according to SLiM-CRAB (S=sixty, Li=light chains, M=MRI, C=calcium [elevated], R=renal failure, A=anemia, B=bone lesions) criteria, myeloma defining events, or date of death, whichever occurs first. As per SLiM-CRAB criteria, clonal bone marrow plasma cell percentage >=60%, Involved : uninvolved serum free Li ratio >= 100, >1 focal lesion on MRI studies, calcium elevation: >0.25 millimole per liter (mmol/L) ( >1 milligram per deciliter [mg/dL]) higher than upper limit of normal or >2.75 mmol/L (>11 mg/dL); creatinine clearance <40 milliliter per minute (mL/min) or serum creatinine >177 micromole per liter (µmol/L) (>2 mg/dL); hemoglobin <10 gram per deciliter (g/dL) (<6.5 mmol/L) or >2 g/dL (>1.25 mmol/L) lower than lower limit of normal; 1 or more osteolytic lesions on skeletal radiography, computed tomography (CT), or positron emission tomography-CT (PET-CT).
The percentage of participants with symptomatic multiple myeloma | Up to 7 years
Response to first subsequent multiple myeloma treatment | Up to 7 years
Overall survival rate | Up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (57):
- United States (15):
  - Little Rock, Arkansas
  - Jacksonville, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - Hackensack, New Jersey
  - New York, New York
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Seattle, Washington
- Australia (4):
  - Box Hill
  - Concord
  - Melbourne
  - Woodville South
- Canada (3):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Toronto, Ontario
- Czechia (3):
  - Brno
  - Hradec Králové
  - Prague
- France (5):
  - Lille
  - Nantes
  - Paris
  - Pierre-Bénite
  - Rennes
- Germany (8):
  - Berlin
  - Chemnitz
  - Essen
  - Heidelberg
  - Mainz
  - München
  - Tübingen
  - Würzburg
- Israel (4):
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Tel Aviv
- Netherlands (3):
  - Amsterdam
  - Rotterdam
  - Utrecht
- Russia (4):
  - Nizhny Novgorod
  - Petrozavodsk
  - Ryazan
  - Saint Petersburg
- Turkey (Türkiye) (4):
  - Ankara
  - Antalya
  - Izmir
  - Samsun
- United Kingdom (4):
  - Cardiff
  - Nottingham
  - Southampton
  - Surrey

REFERENCES:
- [Derived] Landgren O, Chari A, Cohen YC, Spencer A, Voorhees PM, Sandhu I, Jenner MW, Smith D, Cavo M, van de Donk NWCJ, Beksac M, Moreau P, Goldschmidt H, Vieyra D, Sha L, Li L, Rousseau E, Dennis R, Carson R, Hofmeister CC. Efficacy and safety of daratumumab in intermediate/high-risk smoldering multiple myeloma: final analysis of CENTAURUS. Blood. 2025 Apr 10;145(15):1658-1669. doi: 10.1182/blood.2024025897. PMID 39652826
- [Derived] Chari A, Munder M, Weisel K, Jenner M, Bygrave C, Petrucci MT, Boccadoro M, Cavo M, van de Donk NWCJ, Turgut M, Demirkan F, Karadogan I, Libby E, Kleiman R, Kuppens S, Bandekar R, Neff T, Heuck C, Qi M, Clemens PL, Goldschmidt H. Evaluation of Cardiac Repolarization in the Randomized Phase 2 Study of Intermediate- or High-Risk Smoldering Multiple Myeloma Patients Treated with Daratumumab Monotherapy. Adv Ther. 2021 Feb;38(2):1328-1341. doi: 10.1007/s12325-020-01601-w. Epub 2021 Jan 20. PMID 33474705
- [Derived] Landgren CO, Chari A, Cohen YC, Spencer A, Voorhees P, Estell JA, Sandhu I, Jenner MW, Williams C, Cavo M, van de Donk NWCJ, Beksac M, Moreau P, Goldschmidt H, Kuppens S, Bandekar R, Clemens PL, Neff T, Heuck C, Qi M, Hofmeister CC. Daratumumab monotherapy for patients with intermediate-risk or high-risk smoldering multiple myeloma: a randomized, open-label, multicenter, phase 2 study (CENTAURUS). Leukemia. 2020 Jul;34(7):1840-1852. doi: 10.1038/s41375-020-0718-z. Epub 2020 Feb 5. PMID 32024950